CLINICAL TRIAL: NCT01938573
Title: A Phase 1-2 Study of Rapamycin and Cisplatin/Gemcitabine for Treatment of Patients With Bladder Cancer
Brief Title: Sirolimus, Cisplatin, and Gemcitabine Hydrochloride in Treating Patients With Bladder Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Bruce Montgomery, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8027; NCI-2013-01614 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 8027 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2013-09-04; First posted 2013-09-10 (Estimated); Results first posted 2017-10-20 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-09

CONDITIONS: Recurrent Bladder Carcinoma; Stage II Bladder Cancer; Stage III Bladder Cancer; Stage IV Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Gemcitabine; Sirolimus; Cystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sirolimus, cisplatin, gemcitabine (Experimental): Sirolimus day -2, cisplatin 70 mg/m2 IV Day 1 and gemcitabine hydrochloride 1000 mg/m2 IV days 1 and 8 every 21 days for 4 cycles followed by cystectomy (surgery)
  Interventions: Drug: Cisplatin; Drug: Gemcitabine Hydrochloride; Drug: Sirolimus; Procedure: Cystectomy

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroamine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemzar
Drug: Sirolimus — Given PO
  Other Names: Rapamune (RAPA); RAPAMYCIN
Procedure: Cystectomy — Undergo cystectomy when appropriate

SUMMARY:
This phase I/II trial studies the side effects and best dose of sirolimus when given together with cisplatin and gemcitabine hydrochloride and to see how well they work in treating patients with bladder cancer. Biological therapies, such as sirolimus, may stimulate or suppress the immune system in different ways and stop tumor cells from growing. Drugs used in chemotherapy, such as cisplatin and gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving sirolimus together with cisplatin and gemcitabine hydrochloride may be an effective treatment for bladder cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define the maximum-tolerated dose (MTD) of sirolimus (rapamycin) combined with gemcitabine hydrochloride and cisplatin (GC). (Phase I)

II. To determine the pathologic complete response rate at cystectomy in patients with localized, muscle invasive carcinoma of the bladder (clinical tumor [T]2-4, node [N]0 or N1). (Phase II)

SECONDARY OBJECTIVES:

I. To assess the response rate to rapamycin combined with GC. (Phase I)

II. To assess effect of rapamycin with GC on deoxyribonucleic acid (DNA) damage surrogates in cancer associated stroma compared to untreated and GC treated stroma. (Phase I)

III. To assess effect of rapamycin with GC on DNA damage surrogates in cancer associated stroma compared to untreated and GC treated stroma. (Phase II)

IV. To assess toxicity of the MTD dose of rapamycin with GC. (Phase II)

OUTLINE: This is a phase I, dose de-escalation study of sirolimus followed by a phase II study.

Patients receive sirolimus orally (PO) two hours before or after grapefruit juice on day -2, cisplatin intravenously (IV) on day 1 and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients undergo cystectomy as clinically appropriate after 1-4 courses of treatment.

After completion of study treatment, patients are followed up for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (ICF) providing agreement to adhere to the dosing schedule, report for all trial visits and authorization, use and release of health and research trial information
* Histologically or cytologically confirmed carcinoma of the bladder of all histologies except neuroendocrine differentiation or squamous cell histology
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 1
* Eligibility for phase 1 and phase 2 components:

  * Phase 1 - clinical T3 or T4 or N1 or M1 cancer which is untreated or previously treated with platinum based therapy with primary tumor still present in the bladder and amenable to sampling before and after treatment, as indicated
  * Phase 2 - clinical T2-4 N0 or N1 untreated with primary tumor still present in the bladder and amenable to sampling before and after treatment, as indicated
* Life expectancy >= 12 weeks
* No prior malignancy is allowed except:

  * Adequately treated basal cell or squamous cell skin cancer or
  * In situ carcinoma of any site or
  * Other adequately treated malignancy for which the patient is currently disease free for at least one year
* Absolute neutrophil count >= 1.5 x 10^9 cells/L
* Hemoglobin (Hgb) >= 9.0 g/dL
* Platelets >= 100,000 x 10^9/L
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) =< 1.5 x upper limit of normal (ULN)
* Bilirubin and total bilirubin levels =< 1.5 x ULN
* Serum creatinine < 1.5 X institutional ULN mg/dL OR glomerular filtration rate (GFR) >= 50 mL/min
* All pre-study labs required for determination of eligibility are to be completed within 30 days prior to day -2 (or the next business day if falls on a weekend or holiday)
* X-rays and/or scans to assess all disease sites are to be completed within 30 days prior to day -2 (or the next business day if falls on a weekend or holiday)

Exclusion Criteria:

* Patients currently receiving active therapy for other neoplastic disorders
* Known parenchymal brain metastasis
* Active or symptomatic viral hepatitis or chronic liver disease
* Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) class II-IV heart disease or cardiac ejection fraction measurement of < 45 % at baseline, if done
* Atrial fibrillation, or other cardiac arrhythmia requiring medical therapy
* Administration of an investigational therapeutic within 30 days of cycle 1, day 1
* Patients with dementia/psychiatric illness/social situations that would limit compliance with study requirements or would prohibit the understanding and/or giving of informed consent
* Patients with medical conditions, which, in the opinion of the investigators, would jeopardize either the patient or the integrity of the data obtained will not be eligible
* Any condition which, in the opinion of the investigator, would preclude participation in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-10; Primary Completion 2016-08-18 (Actual); Study Completion 2016-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Montgomery, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - VA Puget Sound Health Care System, Seattle, Washington
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 2: Sirolimus day -2, cisplatin 70 mg/m2 IV Day 1 and gemcitabine hydrochloride 1000 mg/m2 IV days 1 and 8 every 21 days for 4 cycles followed by cystectomy (surgery)
  Cisplatin: Given IV
  Gemcitabine Hydrochloride: Given IV
  Sirolimus: Given PO
  Cystectomy: Undergo cystectomy when appropriate
- Phase I: Sirolimus 35 mg PO day -2, cisplatin 70 mg/m2 day 1, gemcitabine 1000 mg/m2 days 1 and 8, every 21 days
Period: Overall Study
Arm/Group | Phase 2 | Phase I
Started | 15 | 6
Completed | 13 | 6
Not Completed | 2 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Operation at other hospital | 1 | 0

BASELINE CHARACTERISTICS:
Population: Patients with either metastatic (phase 1) or localized (phase 2) bladder cancer
Arm/Group | Sirolimus, Cisplatin, Gemcitabine
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 69 [51 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Patients With Dose Limiting Toxicity
Description: Safety will be assessed through summaries of adverse events, vital signs, physical examinations, and clinical laboratory test data (including change from baseline).
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1 - Sirolimus, Cisplatin, Gemcitabine: Sirolimus day -2, cisplatin 70 mg/m2 IV Day 1 and gemcitabine hydrochloride 1000 mg/m2 IV days 1 and 8 every 21 days
  Cisplatin: Given IV
  Gemcitabine Hydrochloride: Given IV
  Sirolimus: Given PO
  Cystectomy: Undergo cystectomy when appropriate
Arm/Group | Phase 1 - Sirolimus, Cisplatin, Gemcitabine
Number analyzed (Participants) | 6
Participants | 0

2. Primary Outcome: Percent of Patients With Pathologic Complete Response (Phase II)
Description: The study will follow an optimal two-stage Simon design based on pathologic complete response rate.
Time Frame: 12 weeks
Population: Patients treated in phase 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus, Cisplatin, Gemcitabine
Number analyzed (Participants) | 15
Participants | 4

3. Secondary Outcome: Incidence of Adverse Events Including Any Unfavorable and Unintended Sign, Symptom, Diagnosis, or Disease Temporally Associated With the Use of a Medicinal Product, Whether or Not Related to the Medicinal Product (Phase I and II)
Description: Graded according to the NCI CTCAE version 4.0. Safety will be assessed through summaries of adverse events, vital signs, physical examinations, and clinical laboratory test data (including change from baseline). All adverse events resulting in discontinuation, dose modification, dosing interruption, and/or treatment delay of study drug will also be listed and tabulated by preferred term.
Time Frame: Up to 28 days after completion of study treatment
Measure: Number; unit: Number of events
Arm/Group | Sirolimus, Cisplatin, Gemcitabine
Number analyzed (Participants) | 21
Number of events | 45

ADVERSE EVENTS:
Time Frame: 4 months (neoadjuvant therapy (3 months) and 1 month after completion)
Arm/Group | Sirolimus, Cisplatin, Gemcitabine
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 21/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus, Cisplatin, Gemcitabine (N=21)
Neutropenia (Blood and lymphatic system disorders) | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (8)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Fatigue (General disorders) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No